CLINICAL TRIAL: NCT02305121
Title: A Focused Registry on the Titanium Trochanter Fixation Nail Advanced (TFNAdvanced™) - TFNA System in Patients With Proximal Inter-, Per- or Subtrochanteric Fractures
Brief Title: Focused Registry on the Titanium Trochanter Fixation Nail Advanced (TFNAdvanced™)
Acronym: FR TFNA
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: FR TFNA
Record Dates: First submitted 2014-11-22; First posted 2014-12-02 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Pertrochanteric Fractures of Femur; Intertrochanteric Fractures of the Femur
Keywords: Trochanteric fracture; Nail; Fracture reduction; Antirotation; trochanteric area with diaphyseal extension; trochanteric area with femoral shaft
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: TFNA — All investigated procedures are part of the standard of care treatment. Only the parker mobility score is study-specific. All patients included are followed up from the time point of enrollment until three months after surgery

SUMMARY:
The aim of this project is the prospective data collection of a new device used for trochanteric fractures of the femur. It should be answered how the newly developed implant called Trochanteric Fixation Nailing with anti-rotation feature (TFNA) is performing clinically and radiological in terms of intra- and postoperative complications.

DETAILED DESCRIPTION:
In comparison to previous implants, the TFNA has been improved substantially. Therefore the purpose of this focused registry is to investigate how the newly developed implant called Trochanteric Fixation Nailing with anti-rotation feature (TFNA) is performing clinically and radiologically in terms of surgical technique, intra- and postoperative complications and short term outcome.

All investigated procedures are part of the standard of care treatment. Only the parker mobility score is study-specific. All patients included are followed up from the time point of enrollment until three months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Pertrochanteric femoral fracture (31-A1 and 31-A2), intertrochanteric fracture (31-A3), fracture of the trochanteric area (31-A1/A2/A3) with diaphyseal extension or combined fracture of the trochanteric area and the femoral shaft (32-A/B/C) treated with the TFNA system according to the technique guide
* Ability to understand the content of the patient information / informed consent form
* Willingness and ability to participate in the registry according to the registry plan (RP)
* Signed and dated IRB/EC-approved written informed consent or assent from a family member

Exclusion Criteria:

* Additional acute fracture
* Any not medically managed severe systemic disease
* Recent history of substance abuse (i.e., recreational drugs, alcohol) that would preclude reliable assessment
* Pregnancy or women planning to conceive within the registry period
* Prisoner
* Participation in any other medical device or medicinal product registry within the previous month that could influence the results of the present registry
* Intraoperative decision to use implants other than the devices under investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with per- or intertrochanteric fractures of the femur, fracture of the trochanteric area with diaphyseal extension or combined fractures of the trochanteric area and the femoral shaft.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
The rate of mechanical and surgical complications defined as the number of | up to 3 months
  * cut out and cut through
  * secondary displacement of parts of the implant
  * breakage of the implant
  * iatrogenic fractures
  * surgical revisions
  * acute deep infection

SECONDARY OUTCOMES:
OR time | Intraoperative
  (in min)
Fracture classification Classification | Baseline
  according to AO/OTA Fracture and Dislocation
Parker Mobility Score | up to 3 months
  Evaluation of the mobility
Quality of reduction and implant placement | up to 3 months
  Based on radiographic analysis with focus on the position of the nail tip relative to the femoral canal and the migration of the head neck element

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blauth, Professor, Principal Investigator — Medical University Innsbruck, Department of Trauma Surgery
Locations (2):
- Medical University Innsbruck, Innsbruck, Austria
- Kantonsspital Baselland, Liestal, Switzerland